CLINICAL TRIAL: NCT03734666
Title: Development of a Mindfulness-Based Treatment for the Reduction of Alcohol Use and Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-19630; R34AT009689 (NIH)
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Use; Alcohol Use, Unspecified
Keywords: alcohol drinking; quit smoking
MeSH Terms: conditions — Tobacco Use; Alcohol Drinking | interventions — Ethanol; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Relapse Prevention (Experimental): Participants will receive Mindfulness Based Relapse Prevention (MBRP), an existing substance use treatment, which has been modified to focus explicitly on smoking cessation and reduced alcohol use, creating Mindfulness Based Relapse Prevention - Smoking and Alcohol (MBRP-SA).
  Interventions: Behavioral: Mindfulness Based Relapse Prevention - Smoking and Alcohol
- Cognitive Behavioral Therapy (Active Comparator): Participants will receive Cognitive Behavioral Therapy (CBT) a well-established and commonly used treatment for substance abuse behaviors that utilizes problem solving and coping skills.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention - Smoking and Alcohol — Mindfulness Based Relapse Prevention (MBRP) is a treatment for preventing relapse in addictive disorders that integrates mindfulness meditation with standard relapse prevention practices.
  Other Names: MBRP
  Arms: Mindfulness Based Relapse Prevention
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT) is a form of therapy that aims to help individuals modify problematic emotions, behaviors, and thoughts.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to develop a treatment that can effectively help people reduce their alcohol use and quit smoking.

DETAILED DESCRIPTION:
This study evaluates a mindfulness-based treatment to concurrently target cigarette smoking and alcohol use behaviors in adults.

Aim 1: Modify an existing mindfulness-based treatment to include a focus on smoking cessation and reduced alcohol use.

Aim 2: Evaluate benchmarks regarding the feasibility and acceptability of Mindfulness Based Relapse Prevention -Smoking and Alcohol Use.

Aim 3: Collect and examine descriptive data on proximal and distal variables associated with increased smoking abstinence and reduced drinking.

ELIGIBILITY:
Inclusion Criteria Aim 1:

* 18 years of age or older
* Currently smoking 3 or more cigarettes per day for the past year.
* Carbon monoxide level >/= 8 ppm(parts per million); should carbon monoxide level yield a result less than 8 ppm, participant will be asked to submit a urine sample to determine contine levels and the result must be >/ level 3
* Participant must be motivated to quit smoking and decrease alcohol use within the next 60 days
* If male, consume >/= 5 drinks and if female consume >/= 4 drinks on at least 1 occasion in the past month
* Willing and able to attend the 8 weekly group sessions
* Valid home address in the Tampa Bay area
* Functioning telephone number
* Can speak, read and write in English

Inclusion Criteria Aim 2:

* 18 years of age or older
* Currently smoking 3 or more cigarettes per day for the past year.
* Motivated to quit smoking and decrease alcohol use within the next 60 days
* If male, consumes >/= 5 drinks and if female consumes >/= 4 drinks on at least 1 occasion in the past month
* Willingness and ability to attend 8 weekly video group sessions
* Willingness and ability to use an email account for study materials
* Valid address
* Functioning telephone number
* Can speak, read and write in English

Exclusion Criteria:

* Unable to wear nicotine patch
* Participants who have an active substance use disorder other than an alcohol use disorder
* Participants who have an active psychotic disorder
* Current use of tobacco cessation medications
* Pregnant or nursing
* Participants who have a household member already enrolled in the study.
* In rare cases, study staff might exclude a participant for a reason not specified here

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Vinci, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vinci C, Sutton SK, Yang MJ, Baban S, Sauls R, Witkiewitz K, Brandon KO, Unrod M, Brandon TH, Wetter DW. Pilot randomized controlled trial of mindfulness-based relapse prevention vs cognitive behavioral therapy for smoking and alcohol use. Drug Alcohol Depend. 2023 Mar 1;244:109768. doi: 10.1016/j.drugalcdep.2023.109768. Epub 2023 Jan 11. PMID 36645978

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
Started | 35 | 32
Completed | 16 | 16
Not Completed | 19 | 16
Not completed — Other | 7 | 4
Not completed — Lost to Follow-up | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 35 | 32 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (9.8) | 43.3 (9.3) | 44.1 (9.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 11 | 9 | 20
  Female | 23 | 23 | 46
  Transgender Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 31 | 28 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 23 | 20 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 35 | 32 | 67

OUTCOME MEASURES:

1. Primary Outcome: Aim 2: Number of Participants Scoring >3
Description: Number of participants scoring >3. Patient satisfaction will be determined through a score on the Client Satisfaction Questionnaire Version 8 (Attkinson & Greenfield), where participants respond to 8 items on a 4-point scale (1=very dissatisfied; 4=very satisfied). Results reported indicate clients with a patient satisfaction score over 80%.
Time Frame: End of Treatment at 8 Weeks
Population: Number of participants analyzed who responded to the survey
Measure: Number; unit: participants
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
Number analyzed (Participants) | 19 | 16
participants | 18 | 16

2. Primary Outcome: Aim 2: Rate of Recruitment of Eligible Participants
Description: Rate of recruitment was measured by calculating the average of eligible participants who were recruited per week
Time Frame: 20 weeks
Measure: Number; unit: participants recruited per week
Groups:
- Eligilible Recruited Participants: Participants were mainly recruited via Trialfacts (a recruitment company that utilized online ads, primarily Facebook and Google ads) and Craigslist ads in Florida and Georgia.
Arm/Group | Eligilible Recruited Participants
Number analyzed (Participants) | 121
participants recruited per week | 6

3. Primary Outcome: Aim 2: Participant Retention
Description: Percentage of participants retained through follow-up
Time Frame: End of study at Week 16 Follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
Number analyzed (Participants) | 35 | 32
percentage of participants | 46 | 50

4. Primary Outcome: Aim 2: Percentage of Participants That Completed Questionnaires
Description: Percentage of participants who completed questionnaires at week 16
Time Frame: End of study at Week 16 Follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
Number analyzed (Participants) | 35 | 32
percentage of participants | 34.7 | 31.4

5. Secondary Outcome: Aim 3: Percent of Smoking Abstinence End of Treatment
Description: Participants will self-report of no smoking in the last 7 days using the 7-day point prevalence.
Time Frame: End of Treatment at 8 Weeks
Population: Non-responders assumed to be smoking
Measure: Number; unit: percentage of participants
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
Number analyzed (Participants) | 35 | 32
percentage of participants | 34.3 | 31.3

6. Secondary Outcome: Aim 3: Percent of Smoking Abstinence at 16 Week Follow-up
Description: Percent of smoking abstinence, measured by biochemical verification of abstinence via saliva continine and self-report of no smoking in the past 7 days. Participants who report abstinence will be mailed a saliva continine kit to confirm abstinence at their 16 week follow up call.
Time Frame: At 16 week follow-up
Population: Non-responders assumed to be smoking
Measure: Number; unit: percentage of participants
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
Number analyzed (Participants) | 35 | 32
percentage of participants | 14.3 | 3.1

7. Secondary Outcome: Aim 3: Percent of Heavy Alcohol Use at End of Treatment
Description: Percent of heavy drinking days during the prior week. Heavy drinking is defined as greater or equal to 4 drinks per day for women and greater or equal to 5 drinks per day for men.
Time Frame: End of Treatment at 8 Weeks
Measure: Mean (Full Range); unit: percentage of heavy drinking days
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
Number analyzed (Participants) | 18 | 16
percentage of heavy drinking days | 4 [0 to 100] | 6.3 [0 to 100]

8. Secondary Outcome: Aim 3: Percentage of Heavy Alcohol Use at 16 Week Follow-up
Description: as for outcome 7
Time Frame: At 16 week follow-up
Measure: Mean (Full Range); unit: percentage of heavy drinking days
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
Number analyzed (Participants) | 16 | 14
percentage of heavy drinking days | 5.1 [0 to 100] | 4.6 [0 to 100]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from start of treatment to end of treatment, an average of 16 weeks.
Arm/Group | Mindfulness Based Relapse Prevention | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/35 | 3/32
Other Adverse Events (participants affected / at risk) | 1/35 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Relapse Prevention (N=35) | Cognitive Behavioral Therapy (N=32)
General Disorders and administration site conditions - Other (General disorders) | 1 (1) | 0 (0) — Participant was admitted to hospital, but did not disclose why
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Torn Ligament (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Relapse Prevention (N=35) | Cognitive Behavioral Therapy (N=32)
Pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03734666/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03734666/ICF_001.pdf